CLINICAL TRIAL: NCT04402788
Title: RAndomized Phase II/III Trial of Consolidation Radiation + Immunotherapy for ES-SCLC: RAPTOR Trial
Brief Title: Testing the Addition of Radiation Therapy to the Usual Immune Therapy Treatment (Atezolizumab) for Extensive Stage Small Cell Lung Cancer, The RAPTOR Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03472; NCI-2020-03472 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU007 (Other: NRG Oncology); NRG-LU007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma
MeSH Terms: interventions — atezolizumab; Specimen Handling; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (atezolizumab) (Active Comparator): Patients receive atezolizumab IV over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT scan, CT, and MRI throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm II (atezolizumab, radiation therapy) (Experimental): Patients receive atezolizumab IV over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy QD on days 1-5 during weeks 1-5 only. Patients undergo PET/CT scan, CT, and MRI throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood and tissue collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm II (atezolizumab, radiation therapy)

SUMMARY:
This phase II/III trial compares the effect of adding radiation therapy to the usual maintenance therapy with atezolizumab versus atezolizumab alone in patients who have already received atezolizumab plus chemotherapy for the treatment of small cell lung cancer that has spread outside of the lung or to other parts of the body (extensive stage). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radiation therapy in addition to atezolizumab may extend the time without extensive small cell lung cancer growing or spreading compared to atezolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare investigator-assessed progression free survival (PFS) between atezolizumab plus radiotherapy and atezolizumab alone. (Phase II) II. To compare overall survival (OS) between atezolizumab plus radiotherapy and atezolizumab alone. (Phase III)

SECONDARY OBJECTIVES:

I. To assess the toxicity between the atezolizumab plus radiotherapy arm and the atezolizumab arm.

II. To assess the impact of adding radiotherapy on PFS and OS in patients with 1-3 visible tumors and > 3 visible tumors.

III. To assess the impact of adding radiotherapy on PFS and OS in patients receiving consolidation radiotherapy to all visible disease ("complete consolidation") and patients who do not receive consolidation radiation to all visible disease ("incomplete consolidation").

EXPLORATORY OBJECTIVE:

I. To assess the association between pre-treatment tumor burden (determined by central radiographic assessment, using both tumor number and tumor volume), and PFS and OS benefit.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive atezolizumab intravenously (IV) over 30 minutes +/- 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive atezolizumab IV over 30 minutes +/- 10 minutes. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy once daily (QD) on days 1-5 during weeks 1-5 only.

Patients undergo positron emission tomography and computed tomography (PET/CT) scan, computed tomography (CT), and magnetic resonance imaging (MRI) throughout the trial. Patients also undergo blood and tissue collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any confirmation (cytologic, histologic, or pathologic) of extensive stage small cell lung cancer at any site, either primary or metastases
* Partial response (PR) or stable disease (SD) after 4-6 cycles of etoposide/platinum (E/P) doublet plus atezolizumab by re-staging scans (positron emission tomography [PET]/computed tomography [CT] scan, diagnostic CT scan, magnetic resonance imaging [MRI] optional per treating physician); atezolizumab should continue through randomization. Patients must be randomized within 9 weeks of last dose of etoposide/platinum (if not receiving PCI) or 6 weeks from completion of prophylactic cranial irradiation (PCI)

  * NOTE: Patients must have at least 3 cycles of E/P plus atezolizumab. They can have one cycle of induction E/P without concurrent atezolizumab if unable to receive concurrent E/P combined with atezolizumab for all cycles of induction therapy
* Patients must have measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST]) and 3 or fewer observable liver metastases and no evidence of progressive disease (per RECIST) at time of enrollment
* At time of enrollment after induction E/P chemotherapy and atezolizumab, if there is a pleural effusion, patients will be eligible if thoracentesis is cytologically negative or if pleural fluid is too small a volume to effectively sample by thoracentesis and does not show increased metabolic activity on CT/PET imaging
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 14 days prior to registration;
  * Imaging within 42 days prior to registration to include:

    * MRI brain with contrast or CT brain with contrast
    * CT chest, abdomen and pelvis or whole body PET/CT scan any time after the fourth cycle of chemotherapy and prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 14 days prior to registration
* Absolute neutrophil count (ANC) >= 1,000/cells/mm^3 (within 14 days prior to registration)
* Platelets >= 75,000 cells/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 8 g/dL (within 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x ULN (AST and/or ALT =< 5 ULN for patients with liver involvement) (within 14 days prior to registration)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 ULN for patients with documented liver involvement or bone metastases) (within 14 days prior to registration)
* Adequate renal function = Creatinine clearance >=40 mL/min by the Cockcroft-Gault (C-G) equation: (within 14 days prior to registration)
* Upfront radiation therapy of symptomatic metastatic site is permissible if causing symptoms such as pain or impending fracture
* Patients with brain metastases are eligible after receiving whole brain radiation before enrollment (anytime during induction systemic therapy). Whole brain radiation can be delivered with hippocampal sparing or 3-D conformal technique. Patients with irradiated brain metastases are eligible if they are clinically stable from a neurological standpoint after completing radiotherapy (e.g. not having uncontrolled seizures) and do not require use of steroids above a dose of 10 mg of prednisone daily
* For women of childbearing potential, a negative serum or urine pregnancy test within 14 days prior to registration.

  * Note: Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patients positive for human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months and a stable regimen of highly active anti-retroviral (HAART) HIV-positive patients must have no requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Metastatic disease invading the liver (> 3 metastases), heart or > 10 metastatic sites detectable after induction systemic therapy. Each visible bone metastasis on radiographic scan counts as one site
* Patients with a concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen with atezolizumab or radiation
* Prior radiotherapy in the thorax that would result in overlapping RT fields, unless the overlapping fields meet acceptable dose constraints for normal tissue
* Active autoimmune disease, including, but not limited to: systemic lupus erythematosus; rheumatoid arthritis; inflammatory bowel disease (e.g. Crohn's, ulcerative colitis); vascular thrombosis associated with antiphospholipid syndrome; Wegener's granulomatosis; Sjogren's syndrome; Guillain-Barre syndrome; multiple sclerosis; vasculitis; or glomerulonephritis.

  * If the autoimmune disease is not active for over 3 years and the patient is not receiving immunosuppressive treatment such as methotrexate or steroids above a dose equivalent to 10 mg prednisone daily, the patient is eligible.
  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations are excluded only if they have active disease with acute exacerbation and on immunosuppressive medications within the 12 months prior to enrollment. They are eligible otherwise.
* Severe, active co-morbidity defined as follows:

  * Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications;
  * Active tuberculosis;
  * Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

    * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). (The HCV RNA test must be performed for patients who have a positive HCV antibody test)
  * Known immunosuppressive disease, for example history of bone marrow transplant or chronic lymphocytic leukemia (CLL);
  * Chronic obstructive pulmonary disease (COPD) requiring chronic oral steroid therapy of > 10 mg prednisone daily or equivalent at the time of registration. Inhaled corticosteroids are not exclusionary;
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months;
  * History of recent myocardial infarction within 6 months prior to registration.
  * Clinically significant interstitial lung disease
* Pregnancy: Administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 5 months (150 days) after the last dose of study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Women who are breastfeeding and unwilling to discontinue
* History of allogeneic organ transplant
* Patients who have had immunotherapy-induced pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Phase II) | From randomization to any documented progression or death due to any cause, whichever occurs first, assessed up to 6 years
  Will compare the distributions of PFS between treatment arms using a one-sided stratified log-rank test in all randomized eligible patients. The rates at various timepoints (e.g., every 6 months after randomization) and medians of PFS for each arm will be estimated using the Kaplan-Meier method. The associated 95% confidence interval (CI) will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Results from an unstratified analysis will also be provided.
Overall survival (OS) (Phase III) | From randomization to the date of death due to any cause, assessed up to 6 years
  Will compare arm I to arm 2 based on OS using a stratified log-rank test. Hazard ratios will be estimated using a stratified Cox regression model. Event rates over time will be estimated within each treatment group using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 years
  For each patient, the maximum severity reported for both immune mediated and non-immune mediated adverse events will be used in the summaries. Adverse events will be summarized regardless of relationship to protocol treatment as assessed by the investigator. All adverse events, adverse events leading to withdrawal, interruption or modification of protocol treatment, grade >= 3 adverse events, and serious adverse events will be summarized. Deaths and cause of death will be summarized. The rate of treatment-related adverse events using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version [v.]5.0) will be reported with the frequency and severity (e.g., type, grade, and attribution) by arm, the analysis will be performed at the time of both phase II and phase III (if applicable) primary endpoint analyses. All adverse events will be classified as either immune or non-immune mediated.
PFS (Phase III) | Up to 6 years
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST). Will compare the distributions of PFS between treatment arms using a one-sided stratified log-rank test in all randomized eligible patients at 0.025 level. The rates at various timepoints (e.g., every 6 months after randomization) and medians of PFS for each arm will be estimated using the Kaplan-Meier method. The associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. If one stratum has less than 10 events, the stratification factor which contains the level with the smallest number of patients will be removed from the stratified analyses.
PFS in patients with 1-3 distinct visible tumors and > 3 distinct visible tumors | Up to 6 years
  Will be similarly summarized and compared between experimental and control. The interaction between the treatment groups and tumor number groups will also be explored in Cox regression model.
OS in patients with 1-3 distinct visible tumors and > 3 distinct visible tumors | Up to 6 years
  Will be similarly summarized and compared between experimental and control. The interaction between the treatment groups and tumor number groups will also be explored in Cox regression model.
PFS in patients receiving consolidation radiotherapy to all visible disease and patients who do not receive consolidation radiotherapy to all visible disease | Up to 6 years
OS in patients receiving consolidation radiotherapy to all visible disease and patients who do not receive consolidation radiotherapy to all visible disease | Up to 6 years

OTHER OUTCOMES:
Tumor burden | Up to 6 years
  Tumor burden determined by central radiographic assessment, using both tumor number and tumor volume will be associated with PFS and OS benefit. The PFS and OS will be similarly summarized and compared between experimental and control in the following subgroups: 1) high or low tumor burden, using >= 4, 5, or 6 metastases as a cutoff; 2) high or low tumor burden, using the median of centrally reviewed radiographic tumor volume as a cutoff.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Nhu Nguyen, Principal Investigator — NRG Oncology
Locations (415):
- United States (415):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Sands Cancer Center, Canandaigua, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Levine Cancer Institute - Union West, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm